CLINICAL TRIAL: NCT00102466
Title: Vildagliptin Compared to Gliclazide in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2338
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Gliclazide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin; Drug: Metformin
- Gliclazide (Active Comparator)
  Interventions: Drug: Gliclazide; Drug: Metformin

INTERVENTIONS:
Drug: vildagliptin
  Arms: Vildagliptin
Drug: Gliclazide
  Arms: Gliclazide
Drug: Metformin

SUMMARY:
This study is not being conducted in the United States. Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to that of gliclazide in lowering overall blood glucose levels when added to metformin in people with type 2 diabetes not at target blood glucose levels on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* On a stable dose of metformin as defined by the protocol
* Blood glucose criteria must be met
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of significant diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 52 weeks | 52 weeks

SECONDARY OUTCOMES:
Adverse event profile after 52 weeks of treatment | 52 weeks
Change from baseline in fasting plasma glucose at 52 weeks | 52 weeks
Patients with endpoint HbA1c <7% at 52 weeks | 52 weeks
Patients with reduction in HbA1c >/= 0.7% after 52 weeks | 52 weeks
Patients with reduction in HbA1c >/= 0.5% after 52 weeks | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Nuremberg, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- See also: Results for CLAF237A2338 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2851